CLINICAL TRIAL: NCT00058487
Title: A Phase II Study Of Epirubicin And Thalidomide In Unresectable Or Metastatic Hepatocellular Carcinoma
Brief Title: Epirubicin and Thalidomide in Treating Patients With Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: DFCI-01281; CDR0000298783 (Registry Identifier: PDQ (Physician Data Query)); CELGENE-2001-P-00170/1
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2006-10

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Epirubicin; Thalidomide

INTERVENTIONS:
Drug: epirubicin hydrochloride
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as epirubicin use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of hepatocellular (liver) cancer by stopping blood flow to the tumor. Combining epirubicin with thalidomide may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining epirubicin with thalidomide in treating patients who have unresectable or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of epirubicin and thalidomide in patients with locally unresectable or metastatic hepatocellular carcinoma.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: Patients receive epirubicin on days 1, 8, and 15 and thalidomide on days 1-21. Courses repeat every 28 days.

PROJECTED ACCRUAL: A total of 12 patients per year will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma

  * Locally unresectable or metastatic disease
* Measurable disease
* No clinically apparent CNS metastases
* No carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 75,000/mm^3

Hepatic

* SGOT no greater than 5 times upper limit of normal
* Bilirubin no greater than 3.0 mg/dL
* INR no greater than 1.5*
* Albumin at least 2.0 g/dL NOTE: *Not required for patients receiving full anticoagulation with warfarin for deep vein thrombosis or pulmonary embolism

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* LVEF normal by echocardiogram or MUGA

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Willing and able to participate in the System for Thalidomide Education and Prescribing Safety (STEPS) program
* No uncontrolled serious medical or psychiatric illness
* No other concurrent uncontrolled malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No more than 1 prior chemotherapy regimen for hepatocellular carcinoma
* No prior chemoembolization to the liver

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* More than 2 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2001-12; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Antitumor activity
Toxic effects

CONTACTS AND LOCATIONS:
Overall Officials: Andrew X. Zhu, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Zhu AX, Fuchs CS, Clark JW, Muzikansky A, Taylor K, Sheehan S, Tam K, Yung E, Kulke MH, Ryan DP. A phase II study of epirubicin and thalidomide in unresectable or metastatic hepatocellular carcinoma. Oncologist. 2005 Jun-Jul;10(6):392-8. doi: 10.1634/theoncologist.10-6-392. PMID 15967833